CLINICAL TRIAL: NCT06673797
Title: Effects of Swiss Ball vs Frenkle Exercises on Static and Dynamic Balance in Ataxic Children With Cerebral Palsy
Brief Title: Effects of Swiss Ball vs Frenkle Exercises on Static and Dynamic Balance in Ataxic CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/Ali Raza
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Ataxic; Balance; Pediatric balance scale; Swiss ball; Frenkel
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be randomized controlled trial in which non probability convenient sampling will be used two groups of ages 5-8 age will be formed in which participants will be randomly divided group A will be receive effects of swiss ball exercises and group B will receive Frenkel exercises on both dynamic and static balance.
Who Masked: Participant
Masking Description: Participant will get separate treatment protocol and possible efforts will be put to mask the both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:The first intervention group would participate in Swiss ball exercises along with stretching (Experimental): Group A: The first intervention group would participate in Swiss ball exercises along with stretching as baseline treatment. The exercises would be performed 3 times per week for four weeks. (12)
  1. Stretching of hamstrings, calf, and quads for 10 seconds hold 5 times. (11)
     1. Calf stretching
     2. Hamstring stretches
     3. Quad stretchings
  2. 2. Swiss ball exercises
     1. Sitting on the Swiss ball with the trunk straight, arms by the sides, and eyes opened progressed towards eyes closed for 10 seconds, then rest
     2. Sitting on the Swiss ball with trunk straight and arm by the sides.
     3. Standing with gym ball in front.
     4. One leg weight bearing on a gym ball with the therapist behind the patient, gripping the patient's pelvis to provide support
  Interventions: Other: Effects of Swiss Ball exercises
- Group B: The second intervention group would participate in Frenkel Exercises along with stretching. (Experimental): 1. Stretching of hamstrings, calf, and quads for 10 seconds hold 5 times. (11)
     1. Calf stretching
     2. Hamstring stretches
     3. Quads stretching
  2. Frenkel's lower limb exercises are the exercises listed below. The time of each session was set to be 10 minutes in the first week and then raised by 5 minutes every week. The patients were given 5 minutes to relax after 10 minutes of practice.
     a. Supine lying: i. with the head lifted; Hip abduction and adduction ii. with the head lifted, and one hip and knee extended iii. with the head lifted; and extending one leg to position the heel on the designated spot b. While sitting: i. stretch one leg to the side, bringing the heel to a spot where a mark has been made on the floor.
     ii. Stride sitting; Stand up from a seated position, then return to a seated position.
     c. Stride standing: i. weight transfer from foot to foot. ii. stepping sideways with feet on floor markings. iii. turn around. iv. walking and turning to avoid obstacles.
  Interventions: Other: EFFECTS OF FRENKEL EXERCISES ON STATIC AND DYNAMIC BALANCE IN ATAXIC CHILDREN WITH CEREBRAL PALSY

INTERVENTIONS:
Other: Effects of Swiss Ball exercises — Effects of Swiss ball exercises along with stretching as baseline treatment.
  1. Stretching of hamstrings, calf, and quads for 10 seconds hold 5 times.
  2. Swiss ball exercises. a.Sitting on the Swiss ball with the trunk straight, arms by the sides, and eyes opened progressed towards eyes closed for 10 seconds, then rest. b.Sitting on the Swiss ball with trunk straight and arm by the sides. The therapist would assist the patient to engage the patient in shifting the body's weight to one side and the other side sideways as well as anterior and posterior and up and down alternatively. Start with 10 repetitions. c. Standing with gym ball in front. The therapist would stand behind the patient to provide support and ask the patient to lean forward on the gym ball with both hands via outstretched arms. Start with 10 repetitions d. One leg weight bearing on a gym ball with the therapist behind the patient, gripping the patient's pelvis to provide support. Start with 10 repetitions
  Arms: Group A:The first intervention group would participate in Swiss ball exercises along with stretching
Other: EFFECTS OF FRENKEL EXERCISES ON STATIC AND DYNAMIC BALANCE IN ATAXIC CHILDREN WITH CEREBRAL PALSY — Frenkel Exercises along with stretching as baseline treatment. The second intervention group would participate in Frenkel Exercises along with stretching as baseline treatment. The exercises would be performed 3 times per week for four weeks.
  1. Stretching of hamstrings, calf, and quads for 10 seconds hold 5 times. (11)
     a. Calf stretching. b. Hamstring stretches. c. Quads stretching
  2. Frenkel's lower limb exercises are the exercises listed below. The time of each session was set to be 10 minutes in the first week and then raised by 5 minutes every week. The patients were given 5 minutes to relax after 10 minutes of practice. (12)
     1. Supine lying
     2. While sitting
     3. Stride standing
  Arms: Group B: The second intervention group would participate in Frenkel Exercises along with stretching.

SUMMARY:
Several studies have highlighted the significant impact of cerebral palsy, a prevailing neurological and musculoskeletal developmental disorder among childhood disabilities worldwide. Within the spectrum of cerebral palsy, ataxic CP stands as the least prevalent type, accounting for 5 to 10% of all cases. Individuals diagnosed with ataxic CP encounter difficulties in fine motor skills, precision, and coordination, and exhibit an unsteady gait, some of which are linked to compromised postural control and inadequate core stability. These issues culminate in functional limitations, heightening the risk of falls, and further contributing to the overall disability experienced by the patients. Consequently, there exists a need to prioritize research and develop targeted treatment protocols specifically for ataxic CP. It is crucial to emphasize the enhancement of postural control and coordination, with particular emphasis on improving static and dynamic balance during rehabilitation. Implementing Swiss ball exercises and Frenkel exercises in the rehabilitation protocol for children with ataxic cerebral palsy can significantly diversify treatment strategies. These exercises play a pivotal role in supporting these children to either sustain or regain their ability to function independently, reduce the risk of falls, and notably improve their overall well-being.

DETAILED DESCRIPTION:
A four-week randomized clinical trial will involve 18 participants, divided randomly into two intervention groups, with nine participants in each group. Group A (intervention group 1) will participate in Swiss ball exercises combined with stretching, while Group B (intervention group 2) will partake in Frenkel exercises along with stretching. The sampling method employed will be a non-probability technique. The Pediatric Balance Scale (PBS) will serve as the primary tool for outcome measurement. Randomization will be conducted using computer-generated software. The study design will be single-blinded, ensuring the assessor remains unaware of the groups' assignments. Initial data collection (pretest) will occur at week 0, followed by post-test data collection at week 4. For intergroup analysis, if the data follows a normal distribution, the parametric Independent t-test will be utilized, enabling the calculation of mean, standard deviation, and p-values. Alternatively, if the data does not display a normal distribution, the non-parametric Mann-Whitney test will be employed, allowing the calculation of median, interquartile ranges, and p-values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with having diagnosis of ataxic cerebral palsy
* Age between 5 to 8 years.
* GMFC level 2.
* Both the genders were included

Exclusion Criteria:

* Visual Impairments and hearing loss
* Mental retardation
* Fixed contractures or deformities of the spine or extremities
* Meningitis

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-11-24 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Pediatric balance scale(PBS) | 15 to 20 minutes
  • Pediatric balance scale (PBS): It is a modified version of the Berg Balance Scale that is used to assess functional (static and dynamic) balance skills before and after exercises in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points. The PBS has a test-retest reliability of ICC=0.998 and a good interrater reliability of ICC=0.997.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Ali Raza Shoukat, MS*, Principal Investigator — Riphah International Univerisity
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pouliot-Laforte A, Parent A, Hamdy R, Marois P, Lemay M, Ballaz L. Relationship between lower limb strength and walking capacities in children with spastic bilateral cerebral palsy. Disabil Rehabil. 2022 May;44(10):1916-1922. doi: 10.1080/09638288.2020.1813819. Epub 2020 Sep 9. PMID 32905745
- [Background] Elshafey MA, Abdrabo MS, Elnaggar RK. Effects of a core stability exercise program on balance and coordination in children with cerebellar ataxic cerebral palsy. J Musculoskelet Neuronal Interact. 2022 Jun 1;22(2):172-178. PMID 35642697